CLINICAL TRIAL: NCT06483464
Title: Validation of the ACS NSQIP Risk Calculator as Predictive Tool for Complications After Thoracic Surgery in Consecutive Series of Patients Operated at the Department of Thoracic Surgery University Hospital Basel
Brief Title: Validation of ACS NSQIP Risk Calculator for Predicting Complications After Thoracic Surgery at University Hospital Basel
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02163; kt24Tsvetkov
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Thoracic
Keywords: Thoracic surgery; Predicting complications; National Surgical Quality Improvement Program of the American College of Surgeons (ACS NSQIP)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single-center retrospective research project aims to evaluate whether and what is the significance of the National Surgical Quality Improvement Program of the American College of Surgeons (ACS NSQIP) risk score in thoracic surgery at the University Hospital Basel.

DETAILED DESCRIPTION:
Advances in medical and surgical therapies have enabled treatment for polymorbid patients, who often have multiple chronic conditions. This has increased the need to accurately assess the risks of postoperative complications and mortality. Due to their complex health status, these patients are more susceptible to adverse outcomes following surgery, necessitating precise risk prediction to guide clinical decision-making and optimize outcomes.

This single-center retrospective research project compares the preoperative risk assessments by the National Surgical Quality Improvement Program of the American College of Surgeons (ACS NSQIP) risk calculator with actual complications (graded according to the Clavien-Dindo classification) observed in patients who underwent thoracic surgery at the University Hospital Basel between May 1, 2021, and March 1, 2022.

The ACS NSQIP risk calculator, a web-based tool, uses 21 preoperative risk factors to predict 13 perioperative outcomes, including serious complications, infections, and mortality. By evaluating these predictions against real patient outcomes, this research project aims to validate the calculator's accuracy specifically in the context of thoracic surgery.

The results of this research project could optimize patient care by better identifying high-risk patients and improving preoperative preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with signed general research consent
* Patients who underwent surgery in our department for the period from 01.05.2021 to 01.03.2022
* Patients with preoperative ACS NSQIP Risk score

Exclusion Criteria:

* Patients who have clearly stated that they would not agree in providing their clinical data for scientific purposes

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A consecutive series of cases of patients who signed the general research consent of the University Hospital Basel and have undergone a thoracic intervention at the University Hospital Basel between 01.05.2021 to 01.03.2022.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Suitability of the ACS NSQIP risk calculator | Up to 30 days after surgery
  To evaluate the suitability of the National Surgical Quality Improvement Program of the American College of Surgeons (ACS NSQIP) risk calculator for thoracic surgery, the ACS NSQIP risk score is compared to actual complications.
  ACS NSQIP risk score is a tool used to predict the likelihood of postoperative complications and mortality in surgical patients. It is calculated based on a range of preoperative variables, including patient demographics, comorbidities, and the type of surgery being performed. The values of the ACS NSQIP risk score can range from 0 to 100, with higher scores indicating a higher risk of complications and a worse expected outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay Tsvetkov, MD, Principal Investigator — Department of Thoracic Surgery, University Hospital of Basel
Locations (1):
- Department of Thoracic Surgery, University Hospital of Basel, Basel, Switzerland